CLINICAL TRIAL: NCT05470062
Title: Effects of Arch Support Insoles on Balance and Gait Performance in Older Adults With Mild Cognitive Impairment
Brief Title: Arch Support Effects on Balance and Gait in Older Adults With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CY Song, Associate professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTH-110-2-5-018
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): wear the insoles for at least 4-h every day for 1-month
  Interventions: Device: arch support insoles (FootDisc)
- control group (No Intervention): not wear insoles for at least 4-h every day for 1-month

INTERVENTIONS:
Device: arch support insoles (FootDisc) — The FootDisc insole is designed with curEVA for shock absorption and motion reduction, poron for secondary heel and metatarsal protection, and dynamic arch support for returning energy for propulsion
  Arms: experimental group

SUMMARY:
This study aims to explore the effects of arch support insoles on balance and gait performance in older adults with mild cognitive impairment (MCI). We will recruit 40 female older adults with MCI. A randomized crossover trial will be used to determine the immediate effect of arch support insoles. All participants received one assessment session wearing and one session not wearing insole in a random order within 1-day. Then participants will be randomly allocated to experimental group (arch support insoles, n=20) or control group (no insoles, n=20) for at least 4-h every day for 1-month. Our primary outcomes include static standing balance, timed-up-and-go test, 10-m obstacle crossing, functional reach test, Short Physical Performance Battery (SPPB), and gait assessment during single- and dual-task walking for 20 m at self-selected comfortable pace while performing serial subtractions (cognitive interference) or carrying a tray (motor interference). Assessments will be conducted at baseline and after 2-wk and 4-wk of insole wear. Statistical analyses will be performed using SPSS 21.0 software. Two-way mixed ANOVA will be used to determine the immediate and short- and long-term effect of arch support insoles. The results of the current study are expected to provide evidences in supporting the use of arch support insoles for improving gait performance and postural stability for older adults with MCI which will contribute to balance and gait training as well as fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* (1) female aged 65 years and over; (2) able to walk more than 20 m without walking aids; (3) had a Montreal Cognitive Assessment (MoCA) score lower than 26 ; (4) had self-reported memory complaints; and (5) had the ability to perform ADLs.

Exclusion Criteria:

* (1) dementia; (2) a history of malignant tumors ; (3) the presence of an unstable neurological or orthopedic disease, or visual problems interfering with participation in the study; and (4) an education level less than 6 years (elementary school).

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of static standing balance | at baseline and after 2-wk and 4-wk of insole wear
  30-s static standing balance
Change of timed-up-and-go test | at baseline and after 2-wk and 4-wk of insole wear
  3-m timed-up-and-go test
Change of 10-m obstacle crossing | at baseline and after 2-wk and 4-wk of insole wear
  10-m obstacle crossing
Change of functional reach test | at baseline and after 2-wk and 4-wk of insole wear
  functional reach test
Change of Short Physical Performance Battery | at baseline and after 2-wk and 4-wk of insole wear
  Short Physical Performance Battery
Change of gait | at baseline and after 2-wk and 4-wk of insole wear
  single- and dual-task walking for 20 m at self-selected comfortable pace while performing serial subtractions (cognitive interference) or carrying a tray (motor interference)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided